CLINICAL TRIAL: NCT02728440
Title: Lipid Profile and Oxidative Stress Parameters of Patients With Idiopathic Hypogonadotropic Hypogonadism and the Change of These Parameters With Gonadotropin Replacement Therapy
Brief Title: Effects of Gonadotropin Replacement Therapy on Metabolic Parameters in Patients With Hypogonadism
Status: Completed | Type: Observational
Sponsor: Gulhane School of Medicine (Other)
Responsible Party: Principal Investigator, Aydogan Aydogdu, MD, Gulhane School of Medicine
Other Study IDs: FB03232016
Record Dates: First submitted 2016-03-27; First posted 2016-04-05 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-03

CONDITIONS: Idiopathic Hypogonadotropic Hypogonadism
MeSH Terms: conditions — Idiopathic Hypogonadotropic Hypogonadism | interventions — Chorionic Gonadotropin; Menotropins

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Hypogonadotropic hypogonadism patients: 30 patients with idiopathic hypogonadotrophic hypogonadism
  Interventions: Drug: human chorionic gonadotropin, human menopausal gonadotropin

INTERVENTIONS:
Drug: human chorionic gonadotropin, human menopausal gonadotropin — drug for the treatment of male hypogonadism
  Other Names: Pregnyl ® Organon hCG 1500 IU; Merional ® ARIS 75 IU

SUMMARY:
Effects of gonadotrophin replacement therapy Lipid Profile and Oxidative Stress Parameters of Patients with Idiopathic Hypogonadotropic Hypogonadism

DETAILED DESCRIPTION:
30 male patients diagnosed with IHH and a control group of 20 healthy cases with similar age and BMI were included in the study. The levels of advanced oxidation protein products (AOPP), thiol, malondialdehyde (MDA), nitric oxide (NO) and 8-hydroxydeoxyguanosine (8-OHdG) and the levels of triglyceride (TG), total cholesterol (TC), high density lipoprotein (HDL-K), low density lipoprotein (LDL-K), Apolipoprotein A1 (ApoA1) and Apolipoprotein B100 (ApoB100) were measured before and after gonadotrophin therapy.

ELIGIBILITY:
Inclusion Criteria:

Serum testosterone concentration < 300ng/dL Absence of a pituitary or hypothalamic mass lesions, Presence of gonadotropin response to GnRH, -

Exclusion Criteria:

diabetes mellitus, arterial hypertension other hormone deficiencies

-

Ages: 22 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with Idiopathic Hypogonadotropic Hypogonadism and healthy control group
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
oxidative stress after hCG and HMG treatment | 2010-2012
HDL levels after hCG treatment | 2010-2012
total cholesterole levels after hCG treatment | 2010-2012

IPD SHARING:
Plan to Share IPD: No